CLINICAL TRIAL: NCT03608826
Title: Relationship Between LINQ™ Subcutaneous Impedance and Right-sided Hemodynamic Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ReLINQuish
Record Dates: First submitted 2018-06-14; First posted 2018-08-01 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm Study (Experimental): Invesigational RAMware will be downloaded onto the LINQ device.
  Interventions: Device: Investigational LINQ™ HF RAMware

INTERVENTIONS:
Device: Investigational LINQ™ HF RAMware — The Reveal LINQ™ device and the 2090 programmer are market-released, but once the investigational LINQ™ HF RAMware is downloaded into the devices, they are considered investigational.

SUMMARY:
The purpose of the ReLINQuish study is to characterize the relationship between subcutaneous impedance and hemodynamic measurements in patients with heart failure. Additionally, the relationship between changes in subcutaneous impedance and other physiologic parameters during acute decompensated HF events will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting at least 1 of 3 criteria will be included in the study:

  * Patients with symptomatic systolic or diastolic heart failure who in the clinician's judgment have a high likelihood of undergoing serial right heart catheterizations to aid in clinical management of their heart failure
  * Patients with dyspnea on exertion in whom exercise hemodynamics is indicated to diagnose diastolic dysfunction
  * Patients who have or will be implanted with a pulmonary artery pressure monitor
* Patient is 18 years of age or older
* Patient (or patient's legally authorized representative) is willing and able to provide written informed consent
* Patient is willing and able to comply with the protocol, including follow-up visits and Carelink transmissions.

Exclusion Criteria:

* Patient has an existing Medtronic implantable cardiac device
* Patient has a left ventricular assist device (LVAD)
* Patient is pregnant (all females of child-bearing potential must have a negative pregnancy test within 1 week of enrollment)
* Patient is enrolled in another study that could confound the results of this study, without documented pre-approval from a Medtronic study manager

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Study: Observational data collection study
Period: Overall Study
Arm/Group | Single Arm Study
Started | 12
Completed | 2
Not Completed | 10
Not completed — Death | 3
Not completed — Heart Transplant | 3
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Study: Single Arm Observational study.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12
History of Coronary Artery Disease [Count of Participants; unit: Participants] | 9
History of Hypertension [Count of Participants; unit: Participants] | 9
History of Atrial Fibrillation [Count of Participants; unit: Participants] | 5
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: %] | 36.0 (21.2)
NYHA class [Count of Participants; unit: Participants] — NYHA Class I-IV with Class I early stage heart failure, and Class IV end stage heart failure.
  Participants
    Class-II | 2
    Class-III | 9
    Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Reveal LINQ™ Subcutaneous Impedance (Units of Ohms) With Pulmonary Artery Pressure (Units of mmHg) From a Swan-Ganz Catheter During Right Heart Catheterization Procedures in Patients With Heart Failure.
Description: The primary objective was to characterize the relationship between changes in Reveal LINQ™ subcutaneous impedance and right heart hemodynamic measurements, resulting from: 1) short-term drug and/or exercise challenges during right heart catheterization procedures or 2) long-term daily trends of physiologic data, in patients with heart failure.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Groups:
- Observation: Observation arm
Arm/Group | Observation
Number analyzed (Participants) | 11
Participants | 0

2. Primary Outcome: Comparison of Reveal LINQ™ Subcutaneous Impedance (Units of Ohms) With Right Atrial Pressure (Units of mmHg) From a Swan-Ganz Catheter During Right Heart Catheterization Procedures in Patients With Heart Failure.
Description: as for outcome 1
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observation
Number analyzed (Participants) | 11
Participants | 0

3. Secondary Outcome: Characterization of the Changes in Reveal LINQ™ Subcutaneous Impedance (Units of Ohms) Prior to Any Acute Decompensated Heart Failure Events.
Description: as for outcome 1
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observation
Number analyzed (Participants) | 9
Participants | 0

4. Secondary Outcome: Characterization of the Changes in Reveal LINQ™ Activity (Units of Hours Per Day) Prior to Any Acute Decompensated Heart Failure Events.
Description: A heart failure event is defined as any cardiovascular-related (including hypervolemia) Health Care Utilizations (HCUs) for any one of the following events.
  * Admission with primary diagnosis of HF
  * Intravenous HF therapy (e.g. IV diuretics/vasodilators) or ultrafiltration at any one of the following settings:
    * Admission with secondary/tertiary diagnosis of HF
    * Emergency Department
    * Ambulance
    * Observation Unit
    * Urgent Care
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observation
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 18 months from enrollment.
Groups:
- Single Arm: Observation Arm
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 3/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=12)
Hospitalization (Cardiac disorders) | 1 — There was one hospitalization which was deemed a serious adverse event on day 285 after insertion procedure which could not be ruled out as related to device or insertion procedure.
Death (Cardiac disorders) | 3

LIMITATIONS AND CAVEATS:
No right heart catheterization was performed during the study, hence the primary outcome could not be summarized. The LINQ device data was not available prior to the acute decompensated heart failure events, hence the secondary outcome could not be summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT03608826/Prot_SAP_000.pdf